CLINICAL TRIAL: NCT04432467
Title: Fertility Restoration Using Autologous Adipose Tissue Derived Mesenchymal Stem Cells
Brief Title: Fertility Restoration Using Autologous Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(Fertility)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Endometritis; Uterus; Scar; Uterine Synechiae; Fallopian Tube Obstruction
Keywords: Fertility restoration; Mesenchymal stem cells
MeSH Terms: conditions — Cicatrix; Gynatresia; Fallopian Tube Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): Patients with impending caesarean section or with chronic inflammation in the mucosa of the uterus and fallopian tubes receiving standard treatment and mesenchymal stem cells
  Interventions: Biological: Autologous mesenchymal stem cells; Other: standard treatment
- control (Active Comparator): Patients with impending caesarean section or with chronic inflammation in the mucosa of the uterus and fallopian tubes receiving standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — Autologous adipose tissue-derived mesenchymal stem cells
  Arms: mesenchymal stem cells
Other: standard treatment — standard treatment according to clinical protocols

SUMMARY:
Treatment of the patients with scarring and adhesions in the uterus resulting from caesarean section or chronic inflammation in the mucosa of the uterus and fallopian tubes and preventing the occurrence of these effects in the future

DETAILED DESCRIPTION:
The aim of the project is to develop a biomedical cell product based on autologous adipose tissue derived mesenchymal stem cells and a biodegradable carrier for highly effective treatment and prevention of scarring and adhesions in the uterus acquired as a result of cesarean section or chronic inflammatory processes in the uterine mucosa and fallopian tubes; to conduct the clinical trials of the biomedical cell product in the treatment of uterus scarring and infertility in women.

ELIGIBILITY:
Inclusion Criteria:

* chronic endometritis
* postoperative uterus scars
* uterine synechia
* fallopian tube obstruction
* absence of acute inflammation in the uterus

Exclusion Criteria:

* Patients with genetic diseases of muscle and connective tissue;
* Patients with malformations of the uterus;
* Acute and chronic infectious diseases: HIV, mycoplasma infection, hepatitis B and C, syphilis; autoimmune diseases; oncological diseases; continuous hormonal therapy with cytostatics corticosteroids; acute noncommunicable diseases;
* mental disorders;
* Drug or alcohol addiction;
* Benign tumors of uterus and appendages;
* Hypersensitivity to any component of the studied biomedical cell product.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 6 months
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  MSC application related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor D Volotovski, Dr, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No